CLINICAL TRIAL: NCT04564430
Title: Clonidine for Tourniquet-related Pain in Children: A Pilot Study
Brief Title: Clonidine for Tourniquet-related Pain in Children
Acronym: CLOTCH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Nicola Groes Clausen, Principle Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NC12547
Record Dates: First submitted 2020-05-25; First posted 2020-09-25 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Polydactyly Toe; Thumb Hypoplasia; Trigger Finger; Polydactyly; Fingers; Osteomyelitis of Hindfoot; Osteomyelitis of Midfoot; Congenital Talipes Equinovarus; Congenital Talipes Calcaneus; Tarsal Coalition; Club Foot; Clubfoot; Congenital Knee Deformity; Leg Length Inequality in Children; Flatfoot; Hollow Foot; Congenital Valgus Foot Deformity; Polydactylia; Polysyndactyly; Syndactyly; Thumb Aplasia; Congenital Hand and Foot Deformity; Subungual Exostosis; Finger Deformity; Toe Deformity; Osteomyelitis of the Foot; Calcaneus Deformity of Foot; Congenital Hand Deformity; Hand Deformities, Congenital; Valgus Foot Deformity; Toe Joint Deformity; Capsulitis of MTP Joint
Keywords: tourniquet; pediatric; clonidine; orthopedic surgery
MeSH Terms: conditions — Thumb deformity; Trigger Finger Disorder; Polydactyly; Clubfoot; Talipes; Tarsal Coalition; Flatfoot; Syndactyly; Foot Deformities; Subungual exostoses; Hand Deformities, Congenital | interventions — Clonidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): IV Saline (Natriumklorid B.Braun 9mg/ml, B.Braun Melsungen AG, Melsungen, Tyskland) in an equal quantity as the study drug is administered at tourniquet inflation
  Interventions: Other: Saline
- Intervention group (Experimental): Catapressan (CatapresR Ampoules 150 micrograms in 1ml, Solution for injection, Boehringer Ingelheim Ltd., Berkshire, UK)(3mcg/kg) is administered at tourniquet inflation
  Interventions: Drug: Catapresan

INTERVENTIONS:
Drug: Catapresan — The intervention is either a single intravenous bolus of 3mcg/kg Catapresan (150mcg/1ml) or an equal amount of saline at the time of tourniquet inflation.
  Other Names: Clonidine
  Arms: Intervention group
Other: Saline — controlgroup receiving saline
  Arms: Control group

SUMMARY:
This study is designed as a randomized, placebo-controlled, double-blinded, clinical trial with two parallel groups.

This study investigates the association between a single dose of the drug, Clonidine, and the total amount of opioid administered under and 24 hours after surgery in children undergoing orthopedic limb surgery with the use of tourniquet.

The investigators hypothesize that administration of clonidine to children undergoing limb surgery with the use of inflatable tourniquets would reduce post-procedural pain.

This study is a pilot to obtain an effect size. Based on this the investigators will calculate a sample size for the main trial enabling us to reach a power of 0.8 with a significans level of 0.05.

DETAILED DESCRIPTION:
Pediatric upper and lower limb surgery often requires fine tissue handling. The prevention of blood flow to a limb allows surgical procedures to be performed with improved accuracy, safety, and speed. Surgical tourniquets, compressing devices used to control venous and arterial circulation to an extremity, enable the surgeons to work in a bloodless operative field.

Tourniquet related complications comprise severe pain during and after the procedure.

In infants and children, surgical procedures are performed under general anaesthesia (GA), comprising standard analgesics and anesthesia maintenance drugs. If an inflatable tourniquet is used, supplementary opioid analgesics are often required to relieve postoperative pain. This clinical observation is in accordance with previously reported data. In adult patients, surgical extremity procedures requiring tourniquets are well known to be painful. As a consequence, infants and children are subjected to prolonged stays in the recovery department. Mobilization and referral to a more child friendly environment might be delayed.

Many interventions and different medications have been tried in order to improve postoperative analgesia in pediatric patients. Amongst these Clonidine, primarily an alpha-2 adrenoceptor agonist. Clonidine stimulates alpha-2 adrenoceptors in the brain stem, thus activating inhibitory neurons, resulting in reduced sympathetic outflow from the CNS.

In several studies' clonidine administered orally or rectally before anesthesia has shown to reduce opioid use and diminish level of pain. Additionally, clonidine reduces the occurrence of postoperative agitation. As an adjuvant to central or peripheral nerve blocks, clonidine effectively prolongs analgesia. The efficacy of clonidine has also been investigated in clinical studies with pediatric ADHD patients Tourette's syndrome and stuttering. The efficacy of Clonidine in these conditions has not been demonstrated.

Clonidine is a taste- and smell less fluid, completely opaque. Although clonidine has been widely studied in the pediatric population, the main outcome of investigations has been emergence delirium. In existing literature, the means of administration vary from intravenous, rectal, epidural or oral dosing. Intravenous single-bolus dosages range from 1.5 - 4 mcg/kg. One recent study included almost 400 patients and administered 3mcg/kg bodyweight without the occurrence of any severe events. Based on these results the investigators chose to administer 3mcg/kg bodyweight as a single bolus in our current study.

All outcomes are objective measures (mg/kg bodyweight, time endurance) or validated evaluation scales (FLACC/VAS score, PAED scale).

Morphine is widely used for postoperative pain relief, the intravenous administration being the most potent. However, morphine is known to have several side effects (prolonged sedation, nausea and vomiting, refusal of oral intake and concomitant dehydration) and may be dangerous for certain children, who experience serious respiratory depression. Hence, a reduction in total dose is crucial, especially after referral to the pediatric ward, where means of monitoring are reduced to intermittent observation and assessment of vital parameters (oxygen saturation by pulse oxymetri, heart rate and blood pressure) is only possible sporadically.

The same is true for pain and the assessment of pain using either FLACC or VAS scales.

Time-at-recovery should be held at a minimum of duration due to high turn-over in our operating facilities. Any unnecessary prolongation of recovery-time should hence be avoided.

Assessment of both primary and secondary outcomes are part of standard care and documentation of the conductance of anesthesia, recovery and post-recovery treatment at the pediatric ward. Hence, this information is readily available but will be registered in source-data sheets. After the individual participant has completed the study, the total amount of morphine administered at the pediatric ward from TREC-END to T24 will be registered by the study investigators.

Prior to any kind of scheduled surgery, patients are seen at the outpatient's clinics at the Department of Orthopedic Surgery. If the patient is less than 15 years of age and is planned for extremity surgery with the use of surgical tourniquet, the surgeon will hand out parental information material. Further, he/she will inquire, whether parents will give their accept to receive a phone call 1-3 days prior to the date of surgery. If parents approve, study investigators will contact the parents and inform them about the study.

If parents agree to study participation, a written consent form will be presented on the day of surgery by one of the study investigators for the parents to sign before induction of anesthesia. Electronic patient records will not be accessed before written consent to study participation has been granted.

All of inclusion- and exclusion criteria are readily available in every anamnesis form filled out in the electronic patient data instrument at Odense University Hospital. Since inclusion criteria comprise 'scheduled procedures', female study participants at fertile ages will hence not be pregnant, since pregnancy is a contraindication against elective/non-urgent surgery with concomitant GA.

On surgery day, children will be prepared according to departmental standard. This includes fasting for meals 6 hours and for watery drinks 1 hour prior to anaesthesia induction and premedication with sedatives at the discretion of the anaesthetist in charge. In order to reduce pre-induction anxiety, parental presence will be allowed and encouraged. Choice of inductional technique (mask or intravenous), choice of airway management device (oral tube (portex (Smiths Medical International Ltd. Bound, Kent, CT21 6JL, UK) or Ruesch (Teleflex Medical, Westmeath, Ireland)) or laryngeal mask (AmbuR AuraStraightTM, Ambu A/S, Ballerup, Denmark) and means of anaesthesia maintenance are according to anaesthetists' preference. After induction, children will receive one i.v. line (BD VenflonTM Pro, Becton Dickinson Infusion Therapy AB, Helsingborg, Sweden) and a bolus of fentanyl (Fentanyl B.Braun; B.Braun Melsungen AG, Melsungen, Tyskland) 3mcg/kg. Maintenance fluid (Ringer's Acetate, Fresenius Kabi AB, Uppsala, Sweden) will be infused at a rate of 10ml/kg the first hour and then reduced to 5ml/kg/h. Monitoring will comprise electrocardiogram (ecg), non-invasive blood pressure (NIBP), puls oxymetri, esohageal temperature (IntelliVue MP70; ViCare Medical, Birkerød, Denmark). Children will be mechanically ventilated by pressure controlled ventilation (Siesta I TS, DAMECA, Denmark) aiming at end tidal carbon dioxide (CO2) of 4.5-5.5kPa. Flow of inspiratory oxygen FiO2 will be set at 45%. Anaesthesia depth will be clinically observed and adjusted as needed. All children will receive paracetamol i.v. (Para15mg/kg after induction. As it is not departmental standard, children will not receive ondansetron or steroid for prophylaxis of post-operative nausea and vomiting (PONV).

Tourniquet will be positioned, and inflation pressure applied according to surgeons' choice. At the time of tourniquet insufflation, children will receive either an intravenous bolus of Catapressan (CatapresR Ampoules 150 micrograms in 1ml, Solution for injection, Boehringer Ingelheim Ltd., Berkshire, UK)(3mcg/kg) or an equal quantity of IV saline (Natriumklorid B.Braun 9mg/ml, B.Braun Melsungen AG, Melsungen, Tyskland). Fentanyl will be supplemented by the anaesthetist as needed according to clinical judgement.

After surgery, children will be awake extubated and transferred to recovery. In recovery, children will be observed and monitored as per departmental standard comprising pulsoxymetri and pain assessment using the FLACC score (<6yrs) and VAS score (>6 yrs). Presence of nausea and vomiting will be registered and treated as per departmental standard. Children will be transferred to the pediatric ward when appropriate, that is in compliance with standards. On the 1st postoperative day the total consumption of opioids 24 hours after transferral to recovery will be summed up.

Peri-anaesthetic data collection: vital parameters (pulse, mean arteria pressure in mmHg, oxygen saturation) will be recorded every 5 minutes. Total amounts in mg/kg of Propofol (intravenous maintenance) or end-tidal sevoflurane/desflurane recorded at time of incision- time of tourniquet inflation and desuflation. Level of tourniquet pressure and total time of insufflation (total-tourniquet-time) will be recorded in minutes. Total amounts of fentanyl (mcg/kg) and infused fluid (ml/kg) will be registered. Adverse events (desaturation <90%, bradycardia and hypotension according to European Pediatric Life Support (EPLS) reference values for age) will be registered.

Recovery: FLACC/VAS score will be recorded at arrival and discharge. If pain is present during recovery, scores will be registered before and after intervention. Total amount of analgesics will be registered. Occurrence of PONV will be registered as well as interventions undertaken against. Occurrence of emergency delirium will be registered. Time-to-discharge will be registered (in minutes).

Children will be transferred to the pediatric ward when appropriate, that is in compliance with standards. On the 1st postoperative day the total consumption of opioids 24 hours after transferral to recovery will be summed up.

The investigators chose the parallel-group design for the CLOTCH-Study. In accordance with ICH-GCP recommendations on statistical principles for clinical trials (E9), the primary analyses will be differences in primary and secondary outcomes adjusted for stratification variables (i.e. means of anaesthesia maintenance (TIVA or Inhalational), tourniquet-time and tourniquet pressure level, age groups <1year, 1-6years, >6years). The investigators will assess and report all outcomes as "intention-to-treat" analysis including all randomised children meeting the inclusion criteria and not fulfilling the exclusion criteria with a standing consent to participate. Complete case analysis will be carried out if the overall level of missing data is less than 5%. However, if exceeding the limit of 5% missing data and if Littles' test is statistically significant, multiple imputation will be used and considered the primary result of the trial to reduce bias from complete case analysis. Little's test tests the null hypothesis that the missing data is Missing Completely At Random (MCAR). A p-value of less than 0.05 is usually interpreted as being that the missing data is not MCAR (i.e. is either Missing At Random or non-ignorable). The investigators will present "worst-case" and "best-case" scenarios. p < 0.05 will be considered statistically significant. For each group, all children will be analysed for the primary outcome. For each primary and secondary outcome, the results and estimated effect sizes with 95% confidence interval will be provided. The investigators will exclude patients with major protocol violations defined as failure to receive the total drug dose. The investigators will carry out statistical analyses before revealing the code of allocation.

The trial offers benefits for the population, which the minor study participant represents. These comprise

* Improved strategies for treatment of pain after use of surgical tourniquets for extremity surgery
* Reduced anxiety and discomfort postoperatively due to reduced pain levels
* Accelerated mobilization postoperatively - a major factor in order to prevent immobility related complications (pulmonary infections, obstipation)
* Reduced-time-to-oral-intake, which is extremely important in all age groups, but crucial for infants, who have a high metabolism and hence are at high risk of complications due to anaerobic energy production.

ELIGIBILITY:
Inclusion Criteria:

* ASA I + II
* Scheduled for GA and planned for relevant surgical procedure (according to table 1)
* Planned use of surgical tourniquet on upper and/or lower extremity

Exclusion Criteria:

* parental consent missing
* ASA classification >II
* Known diagnosis of QT-prolongation syndrome
* known allergies to clonidine
* known allergies or intolerance to morphine
* daily use of pain killers
* under treatment with antihypertensive and antiarrythmic medications
* status of current or previous prematurity
* planned for peripheral or central nerve block in addition to general anaesthesia

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine T24 | Through time spent in the Post-Anaesthesia Care Unit (PACU), i.e. from end-of-incision time to time of transferal from PACU to the paediatric ward, maxium up to 24 hours
  Total amount of i.v. morphine in milligram (mg) administered per kg bodyweight from end-of-incision-time (T0) through the first 24 hours postoperatively (T24).

SECONDARY OUTCOMES:
Morphine recovery to transferal to pediatric ward | Through time spent at the paediatric ward, i.e. from time of transferal from PACU to the paediatric ward to time of discharge up to 24 hours after end-of-incision-time
  Total amount of i.v. morphine in mg administered per kg bodyweight during recovery, i.e. from end-of-incision-time (T0) to time at transferal to the paediatric ward (TREC-END)
Morphine at pediatric ward to T24 | Through time spent in the Post-Anaesthesia Care Unit (PACU), i.e. from end-of-incision time to time of transferal from PACU to the paediatric ward, maximum up to 24 hours
  Total amount of i.v. morphine in mg administered per kg bodyweight in the paediatric ward from time at transferal to the paediatric ward (TREC-END) until 24-hours after end-of-incision-time (T24)
Total time at recovery | Through time spent in the Post-Anaesthesia Care Unit (PACU), i.e. from end-of-incision time to time of transferal from PACU to the paediatric ward, maximum up to 24 hours
  The total time spent in recovery at PACU (TREC-total)
Maximal pain | Through time spent in the Post-Anaesthesia Care Unit (PACU), i.e. from end-of-incision time to time of transferal from PACU to the paediatric ward, maximum up to 24 hours
  For children between the ages of 2 months and 7 years, maximal pain during recovery at PACU will be assessed using the 'Face, Legs, Activity, Cry, Consolability' (FLACC) scale ranging from score 1-10.
  For children above 7 years pain during recovery at PACU was assessed by a Visual Analog Score (VAS) also ranging from 1 to 10.
Occurrence of emergence delirium(ED) | Through time spent in the Post-Anaesthesia Care Unit (PACU), i.e. from end-of-incision time to time of transferal from PACU to the paediatric ward, maximum up to 24 hours
  Occurrence of ED assessed by Paediatric Anaesthesia Emergence Delirium (PAED) scale (1-5). 5 representing highest level of emergence delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola G. Clausen, Ph.D., Principal Investigator — Department of Anaesthesiology and Intensive Care at Odense University Hospital; Tom G. Hansen, Ph.D., Study Director — Department of Anaesthesiology and Intensive Care at Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Budic I, Pavlovic D, Kitic D, Kocic G, Cvetkovic T, Simic D, Jevtovic-Stoimenov T. Tourniquet-induced ischemia-reperfusion injuries during extremity surgery at children's age: impact of anesthetic chemical structure. Redox Rep. 2013;18(1):20-6. doi: 10.1179/1351000212Y.0000000037. PMID 23394494
- [Background] Kumar K, Railton C, Tawfic Q. Tourniquet application during anesthesia: "What we need to know?". J Anaesthesiol Clin Pharmacol. 2016 Oct-Dec;32(4):424-430. doi: 10.4103/0970-9185.168174. PMID 28096570
- [Background] Kruse H, Christensen KP, Moller AM, Gogenur I. Tourniquet use during ankle surgery leads to increased postoperative opioid use. J Clin Anesth. 2015 Aug;27(5):380-4. doi: 10.1016/j.jclinane.2015.03.034. Epub 2015 May 12. PMID 25979462
- [Background] Rudkin AK, Rudkin GE, Dracopoulos GC. Acceptability of ankle tourniquet use in midfoot and forefoot surgery: audit of 1000 cases. Foot Ankle Int. 2004 Nov;25(11):788-94. doi: 10.1177/107110070402501106. PMID 15574237
- [Background] Budic I, Pavlovic D, Kocic G, Cvetkovic T, Simic D, Basic J, Zivanovic D. Biomarkers of oxidative stress and endothelial dysfunction after tourniquet release in children. Physiol Res. 2011;60(Suppl 1):S137-45. doi: 10.33549/physiolres.932170. Epub 2011 Jul 19. PMID 21777032
- [Background] Estebe JP, Davies JM, Richebe P. The pneumatic tourniquet: mechanical, ischaemia-reperfusion and systemic effects. Eur J Anaesthesiol. 2011 Jun;28(6):404-11. doi: 10.1097/EJA.0b013e328346d5a9. PMID 21502865
- [Background] Gourdin M, Dubois P, Mullier F, Chatelain B, Dogne JM, Marchandise B, Jamart J, De Kock M. The effect of clonidine, an alpha-2 adrenergic receptor agonist, on inflammatory response and postischemic endothelium function during early reperfusion in healthy volunteers. J Cardiovasc Pharmacol. 2012 Dec;60(6):553-60. doi: 10.1097/FJC.0b013e31827303fa. PMID 22987052
- [Background] Jellinge ME, Petersen RH. [Clonidine can reduce opioid medication during post-operative pain]. Ugeskr Laeger. 2015 Nov 30;177(49):V05150415. Danish. PMID 26651552
- [Background] Isaac L. Clonidine in the central nervous system: site and mechanism of hypotensive action. J Cardiovasc Pharmacol. 1980;2 Suppl 1:S5-19. PMID 6154837
- [Background] Ydemann M, Nielsen BN, Wetterslev J, Henneberg S, Lauritsen T, Steen N, Edstrom B, Afshari A. Effect of clonidine to prevent agitation in children after sevoflurane anaesthesia: a randomised placebo controlled multicentre trial. Dan Med J. 2016 Jun;63(6):A5234. PMID 27264945
- [Background] Lambert P, Cyna AM, Knight N, Middleton P. Clonidine premedication for postoperative analgesia in children. Cochrane Database Syst Rev. 2014 Jan 28;2014(1):CD009633. doi: 10.1002/14651858.CD009633.pub2. PMID 24470114
- [Background] Boric K, Dosenovic S, Jelicic Kadic A, Batinic M, Cavar M, Urlic M, Markovina N, Puljak L. Interventions for postoperative pain in children: An overview of systematic reviews. Paediatr Anaesth. 2017 Sep;27(9):893-904. doi: 10.1111/pan.13203. Epub 2017 Jul 14. PMID 28707454
- [Background] Wang W, Huang P, Gao W, Cao F, Yi M, Chen L, Guo X. Efficacy and Acceptability of Different Auxiliary Drugs in Pediatric Sevoflurane Anesthesia: A Network Meta-analysis of Mixed Treatment Comparisons. Sci Rep. 2016 Nov 10;6:36553. doi: 10.1038/srep36553. PMID 27830713
- [Background] Moore AD, Anghelescu DL. Emergence Delirium in Pediatric Anesthesia. Paediatr Drugs. 2017 Feb;19(1):11-20. doi: 10.1007/s40272-016-0201-5. PMID 27798810
- [Background] Afshari A. Clonidine in pediatric anesthesia: the new panacea or a drug still looking for an indication? Curr Opin Anaesthesiol. 2019 Jun;32(3):327-333. doi: 10.1097/ACO.0000000000000724. PMID 31045639
- [Background] Ydemann M, Nielsen BN, Henneberg S, Jakobsen JC, Wetterslev J, Lauritsen T, Steen N, Edstrom B, Afshari A; PREVENT AGITATION Research Group. Intraoperative clonidine for prevention of postoperative agitation in children anaesthetised with sevoflurane (PREVENT AGITATION): a randomised, placebo-controlled, double-blind trial. Lancet Child Adolesc Health. 2018 Jan;2(1):15-24. doi: 10.1016/S2352-4642(17)30127-X. Epub 2017 Nov 2. PMID 30169192
- [Background] Khetani JD, Madadi P, Sommer DD, Reddy D, Sistonen J, Ross CJ, Carleton BC, Hayden MR, Koren G. Apnea and oxygen desaturations in children treated with opioids after adenotonsillectomy for obstructive sleep apnea syndrome: a prospective pilot study. Paediatr Drugs. 2012 Dec 1;14(6):411-5. doi: 10.2165/11633570-000000000-00000. PMID 23013460
- [Background] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387
- [Background] Jay MA, Thomas BM, Nandi R, Howard RF. Higher risk of opioid-induced respiratory depression in children with neurodevelopmental disability: a retrospective cohort study of 12 904 patients. Br J Anaesth. 2017 Feb;118(2):239-246. doi: 10.1093/bja/aew403. PMID 28100528
- [Background] Oderda GM, Senagore AJ, Morland K, Iqbal SU, Kugel M, Liu S, Habib AS. Opioid-related respiratory and gastrointestinal adverse events in patients with acute postoperative pain: prevalence, predictors, and burden. J Pain Palliat Care Pharmacother. 2019 Sep-Dec;33(3-4):82-97. doi: 10.1080/15360288.2019.1668902. Epub 2019 Oct 14. PMID 31609155
- [Background] Berghmans JM, Poley MJ, van der Ende J, Weber F, Van de Velde M, Adriaenssens P, Himpe D, Verhulst FC, Utens E. A Visual Analog Scale to assess anxiety in children during anesthesia induction (VAS-I): Results supporting its validity in a sample of day care surgery patients. Paediatr Anaesth. 2017 Sep;27(9):955-961. doi: 10.1111/pan.13206. Epub 2017 Jul 14. PMID 28707384
- [Background] Malviya S, Voepel-Lewis T, Burke C, Merkel S, Tait AR. The revised FLACC observational pain tool: improved reliability and validity for pain assessment in children with cognitive impairment. Paediatr Anaesth. 2006 Mar;16(3):258-65. doi: 10.1111/j.1460-9592.2005.01773.x. PMID 16490089
- [Background] Pedersen LK, Rahbek O, Nikolajsen L, Moller-Madsen B. The revised FLACC score: Reliability and validation for pain assessment in children with cerebral palsy. Scand J Pain. 2015 Oct 1;9(1):57-61. doi: 10.1016/j.sjpain.2015.06.007. PMID 29911640